CLINICAL TRIAL: NCT06332859
Title: Effectiveness of a Resilience-based Rehabilitation Program in Patients with TakoTsubo Cardiomyopathy and After Acute Coronary Syndrome
Brief Title: Effectiveness of a Resilience-Based Rehabilitation Program for Patients with Coronary Heart Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pensionsversicherungsanstalt (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FOR-0022
Record Dates: First submitted 2024-03-20; First posted 2024-03-27 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2024-11

CONDITIONS: Takotsubo Cardiomyopathy; Acute Coronary Syndrome; Psychological Resilience
MeSH Terms: conditions — Takotsubo Cardiomyopathy; Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TakoTsubo (Experimental): Individuals with TakoTsubo cardiomyopathy who participate in an inpatient rehabilitation programme receive an additional psychological intervention, specifically resilience training. This is not a common practice in such rehabilitation programmes.
  Interventions: Other: Resilience training
- Acute coronary event (Experimental): Individuals after an acute coronary event who participate in an inpatient rehabilitation programme receive an additional psychological intervention, specifically resilience training. This is not a common practice in such rehabilitation programmes.
  Interventions: Other: Resilience training

INTERVENTIONS:
Other: Resilience training — The resilience training consists of two sessions of psychological group therapy, each lasting 100 minutes, with a special focus on resilience. Additionally, there are two sessions of relaxation training, known as 'heart yoga', each lasting 25 minutes.

SUMMARY:
To handle daily life challenges, one needs to be psychologically resilient. It plays a crucial role in disease development, prognosis, as well as social, occupational, and community participation. Cardiovascular diseases cause physical and psychological stress, which can be linked to individual resilience and the development of such diseases. Stress can trigger TakoTsubo cardiomyopathy and acute coronary events. Individuals who have experienced TakoTsubo cardiomyopathy or an acute coronary event often feel stressed due to emotional or physical triggers. These triggers may include job loss or illness. In medical rehabilitation, therapists consider the individual circumstances of their patients when planning therapy. It may be important to add a special focus on psychological care, including building resilience, which could greatly benefit these individuals. Therefore, the study aims to investigate whether resilience training, as part of an inpatient multidisciplinary rehabilitation program, affects the individual resilience of rehabilitants with TakoTsubo cardiomyopathy or those who have experienced an acute coronary event.

DETAILED DESCRIPTION:
To cope with the demands of everyday life, individuals require a certain level of psychological resilience. Resilience can be defined in various ways, such as the interplay between vulnerability (risk factors) and protection (resources). Another definition of resilience is the ability to adapt positively to stressful circumstances or to remain functionally stable and healthy despite prolonged stress. Resilience is a crucial factor in determining the quality of life and the psychosocial behaviour of an individual. Therefore, measuring individual resilience can help to understand an individual's resistance to stress and to initiate appropriate therapeutic interventions. There is evidence to suggest that cardiovascular diseases can cause increased physical and psychological stress in patients, potentially indicating a link between individual resilience and cardiovascular disease. Specifically, stress can lead to conditions such as takotsubo cardiomyopathy and acute coronary events. Individuals with takotsubo cardiomyopathy or those who have experienced an acute coronary event often encounter stress as a result of acute emotional or physical triggers, such as job loss or illness. Additionally, those affected often describe long-lasting stress, such as post-traumatic stress disorder or suppression of emotions, before the onset of symptoms.

The symptom complex of takotsubo cardiomyopathy are similar to those of an acute myocardial infarction, but without narrowed coronary arteries. Additionally, takotsubo cardiomyopathy is more prevalent in postmenopausal women. Studies have shown that the mortality rate of takotsubo cardiomyopathy is higher than previously assumed. Additionally, the long-term mortality of patients with takotsubo cardiomyopathy is higher than that of patients after a heart attack.

As medical rehabilitation is a commonly used method for treating cardiovascular diseases. It has been shown to be effective in sustaining the benefits of acute hospital treatment. However, this approach is often overlooked in patients with takotsubo cardiomyopathy, despite its proven positive effects.

A multidisciplinary team can provide individualized care to patients as part of a medical rehabilitation process. The provision of psychological support, such as coping strategies and resilience building, could be of great benefit to people undergoing rehabilitation for takotsubo cardiomyopathy. Research indicates that patients diagnosed with takotsubo cardiomyopathy often struggle to manage stress for an extended period following their diagnosis and initial treatment, which can negatively impact their quality of life and participation. Furthermore, compared to the general population, patients who have been treated for an acute cardiac event, such as an acute myocardial infarction, have lower stress tolerance.

Therefore, the aim of this research project is to assess the effectiveness of a resilience-focused rehabilitation programme for people with takotsubo cardiomyopathy or who have experienced an acute coronary event.

This study will examine changes in psychological resilience, as measured by two independent resilience scales (Resilience Scale-13 and Brief Resilience Scale), during three weeks of inpatient rehabilitation and assess sustainability of these changes after completion of rehabilitation (six-month follow-up). Additionally, participation-related parameters (health-related quality of life, psychological distress and work ability) and physical performance (incremental cycle ergometry) will also be considered.

ELIGIBILITY:
Inclusion Criteria:

* patients experienced TakoTsubo cardiomyopathy (I42.88, I42.9) or patients after an acute coronary event (I21.9) (max. 6 month post event)
* older than 18 years
* signed consent form

Exclusion Criteria:

* Acute intercurrent illness (longer than 3 days)
* No sufficient knowledge of German to enable participation in the resilience training (assessment by recruiting person)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2026-10-14 (Estimated); Study Completion 2026-10-14 (Estimated)

PRIMARY OUTCOMES:
Resilience scale-13 (RS-13) | 3 weeks of inpatient rehabilitation + 6 month follow-up
  The resilience scale-13 measures individual resilience using 13 items on a 7-point Likert scale. The RS-13 scale measures the following aspects of the resilience concept: optimism, emotional stability, zest for life, energy, openness to new things and the ability to change perspective. It can be divided into two factors (competence and acceptance) and describe overall resilience. The scale values range from 1 = "strongly disagree" to 7 = "strongly agree". Higher values meaning higher resilience.
Brief Resilience scale - German Version (BRS) | 3 weeks of inpatient rehabilitation + 6 month follow-up
  The brief resilience scale (German Version) measures the self-assessment of an individual's ability to recover from stress despite considerable adversity. The BSR-D consists of six items. The items are rated on a 5-point likert scale (1 = strongly disagree to 5 = strongly agree). Higher values meaning higher resilience.

SECONDARY OUTCOMES:
European Quality of Life 5 Dimensions 5 Level (EQ-5D-5L) | 3 weeks of inpatient rehabilitation + 6 month follow-up
  The EQ-5D-5L is a general instrument for measuring patient-reported outcomes (PROs), which can be used to assess the quality of life of patients on different dimensions (mobility, self-care, usual activities, pain/discomfort) on a 5-level scale (Min. = 0, Max. = 5). Lower values indicate less impairments in the respective dimensions.
  Moreover, the EQ-5D-5L assesses the patient's self-rated health on a 100 point visual analog scale (Min. = 0, Max. =100). Lower values indicate less positive ratings of health.
Patient Health Questionnaire-4 (PHQ-4) | 3 weeks of inpatient rehabilitation + 6 month follow-up
  The Patient Health Questionnaire-4 (PHQ-4) operationalizes core criteria for anxiety and depression on a 4 point likert scale (Min. = 0, Max = 4). Lower values indicate less impairments.
Maximal incremental exercise test | 3 weeks of inpatient rehabilitation
  The maximal incremental exercise test is performed on a stationary cycle ergometer. The size of the increments is personalized (5-30 watt) for each patient based on their predicted peak work. Increments are increased every minute, allowing the patient to reach peak workload within 8-12 minutes.
Work ability index (WAI) | 3 weeks of inpatient rehabilitation + 6 month follow-up
  The Work Ability Index (WAI) is an instrument for assessing work ability. (Min. = 7, Max = 49). Lower values indicate less subjective work ability.

CONTACTS AND LOCATIONS:
Overall Officials: Doreen Stöhr, Mag., Study Chair — Austrian Pension Insurance Institution
Locations (1):
- Rehabilitationszentrum Bad Tatzmannsdorf, Bad Tatzmannsdorf, Burgenland, Austria

IPD SHARING:
Plan to Share IPD: No